CLINICAL TRIAL: NCT03107377
Title: Phase 2B Double-blind Placebo-controlled Efficacy Trial of EVO100 (Previously Known as Amphora ® Gel) for the Prevention of Acquisition of Urogenital Chlamydia Trachomatis Infection
Brief Title: Phase 2B/3 Double-blinded Placebo-controlled
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Evofem Inc. (Industry)
Collaborators: Clinical Research Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EVO-003
Record Dates: First submitted 2017-03-29; First posted 2017-04-11 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Chlamydia Trachomatis Infection

STUDY DESIGN:
Intervention Model Description: Phase 2B double-blind placebo-controlled efficacy trial of EVO100 for the prevention of acquisition of urogenital Chlamydia trachomatis infection
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind placebo-controlled efficacy trial of EVO100
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EVO100 (Active Comparator): A pH-buffering, acidity-maintaining gel (pH 3.5), containing three active compounds: lactic acid, citric acid, potassium bitartrate. 5 g intravaginally applied at least one hour prior to vaginal intercourse.
  Interventions: Drug: EVO100
- Placebo (Placebo Comparator): An isotonic, non-buffering gel, pH adjusted to 4.5, containing 2.7% hydroxyethylcellulose, sorbic acid, sodium hydroxide, sodium chloride and purified water. 5 g intravaginally applied at least one hour prior to vaginal intercourse.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EVO100 — 5 g dose applied up to 1 hour prior to coitus
  Arms: EVO100
Drug: Placebo — 5 g dose applied up to 1 hour prior to coitus
  Arms: Placebo

SUMMARY:
Phase 2B double-blind placebo-controlled efficacy trial of EVO100 (previously known as Amphora ® Gel) for the prevention of acquisition of urogenital Chlamydia trachomatis infection

DETAILED DESCRIPTION:
Primary: To determine if intravaginal EVO100 reduces the risk of urogenital Chlamydia trachomatis (CT) infection.

Secondary: To determine if intravaginal EVO100 reduces the risk of urogenital Neisseria gonorrhoeae (GC) infection.

Exploratory:To determine if EVO100 use rate (subject adherence to instructed use) has an effect on proportion of subjects who experience CT or GC infection during the study intervention period.

Primary Outcome Measures: Proportion of subjects who experience urogenital CT infection during the study intervention period (incident infection of CT).

Secondary Outcome Measures: Proportion of subjects who experience urogenital GC infection during the study intervention period (incident infection of GC).

Exploratory Outcome Measures:

* Compliance with EVO100 usage during study (rate of product use adherence).
* Sensitivity analyses of the primary parameter (proportion of subjects who experience at least one CT or GC infection during the study intervention period) will be performed for the following:
* Subjects with ≥20%, ≥40%, ≥60% and ≥80% product use adherence
* Subject Satisfaction
* Sexual satisfaction

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects between 18 and 45 years, inclusive
2. Ability to understand the consent process and procedures
3. Subjects agree to be available for all study visits
4. Written informed consent in accordance with institutional guidelines
5. Negative pregnancy test
6. Negative CT and GC NAAT tests OR positive CT or GC NAAT and receives standard of care (SOC) treatment
7. Agree to use a woman-controlled method of contraception, such as oral contraceptives, vaginal ring, birth control implants, IUDs, or tubal ligation (with the exception of spermicides, diaphragms, or any vaginally applied or inserted products containing nonoxynol-9). Condom use only is not an acceptable form of contraception for this study.
8. Able and willing to comply with all study procedures
9. Documented (as part of a retrievable medical record) CT or GC infection within 16 weeks prior to enrollment
10. Reports vaginal sexual intercourse with a male partner at least 3 times per month in the previous month and anticipates vaginal sexual intercourse regularly for the duration of the study
11. Agree to abstain from douching or any form of vaginal suppository use (other than study product) during course of study

    -

Exclusion Criteria:

1. Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
2. In the opinion of the Investigator, have a history of substance abuse in the last 12 months
3. In the opinion of the Investigator, have issues, conditions, or concerns that may compromise the safety of the subject, impact the subject's compliance with the protocol requirements, or confound the reliability of the data acquired
4. Be an Evofem, ClinicalRM, or clinical site employee regardless of direct involvement in research activities, or their close relative
5. Pregnant (or actively trying to become pregnant), or breast-feeding
6. Women who have undergone a total hysterectomy (had uterus and cervix removed)
7. Inability to provide informed consent
8. A subject with a history or expectation of noncompliance with medications or intervention protocol
9. Have engaged in sexual intercourse, douching or used of any form of vaginal suppository or intravaginal device for 24 hours prior to enrollment (may be enrolled at a later date if all other criteria are met)
10. Menstruating at enrollment (may be enrolled at a later date if all other criteria are met)
11. Women who are currently being treated, or have been treated, for a period of 14 days prior to enrollment, with specific antibiotics known to be used for the treatment of CT or GC:

    1. Azithromycin
    2. Erythromycin
    3. Tetracycline
    4. Minocycline
    5. Doxycycline
    6. Levofloxacin
    7. Ofloxacin
    8. Ceftriaxone
    9. Cefixime
12. In the opinion of the Investigator, has signs/symptoms that indicate persistence of chlamydia or gonorrhea infection diagnosed at screening, new interval infection and/or a failure to comply with or complete the prescribed treatment regimen following a positive screening NAAT.
13. Women who regularly use douches, vaginal medications, products, or suppositories
14. Women who are currently using contraceptive products that are directly delivered to the vaginal mucosa, such as diaphragms, vaginal rings (e.g. NuvaRing®), spermicides, or any vaginally applied or inserted products containing nonoxynol-9.
15. Children, pregnant women, prisoners, and other vulnerable populations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 844 female subjects, ages 18-45.
Enrollment: 860 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Culwell, MD, Study Director — Evofem Inc.
Locations (50):
- United States (50):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Mobile OB-GYN, PC, Mobile, Alabama
  - MedPharmics, LLC, Phoenix, Arizona
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - California Center for Clinical Research, Arcadia, California
  - Hope Clinical Research, Canoga Park, California
  - United Clinical Research, Huntington Park, California
  - Medical Center for Clinical Research - Wake Research, San Diego, California
  - Optimus Medical Group, Inc., San Francisco, California
  - AFC Urgent Care Denver, Denver, Colorado
  - Planned Parenthood of Southern New England, New Haven, Connecticut
  - Precision Clinical Research, Lauderdale Lakes, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - Physician Care Clinical Research LLC, Sarasota, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Columbus Regional Research Institute - IACT Health, Columbus, Georgia
  - Renew Health Clinical Research, LLC, Lawrenceville, Georgia
  - Meridian Clinical Research, Richmond Hill, Georgia
  - ASR, LLC, Nampa, Idaho
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - DM Clinical Research, Alexandria, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Valley OB-GYN, Saginaw, Michigan
  - MedPharmics, LLD, Biloxi, Mississippi
  - University of MS Medical Center, Jackson, Mississippi
  - Nevada Obstetrical Charity Clinic, Las Vegas, Nevada
  - Bosque Women's Care, Albuquerque, New Mexico
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research, Inc. - Wilmington Health, Wilmington, North Carolina
  - University of Cincinnati Physicians, Cincinnati, Ohio
  - Planned Parenthood Southeastern Pennsylvania, Philadelphia, Pennsylvania
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Invocare Clinical Research Center, West Columbia, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Adams Patterson OB/GYN, Medical Research Center of Memphis, Memphis, Tennessee
  - Premier Family Physicians, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - CityDoc Urgent Care, Dallas, Texas
  - Research Network America, Houston, Texas
  - Centex Studios, Inc., Houston, Texas
  - Discovery MM Services, Inc., Houston, Texas
  - S.E.Tx. Family Planning and Cancer Screening (SOGA), Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - North Texas Family Medicine, Plano, Texas
  - Neere Bhatia, MD OB/GYN, San Antonio, Texas
  - The Group for Women, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chappell BT, Mena LA, Maximos B, Mollan S, Culwell K, Howard B. EVO100 prevents chlamydia and gonorrhea in women at high risk of infection. Am J Obstet Gynecol. 2021 Aug;225(2):162.e1-162.e14. doi: 10.1016/j.ajog.2021.03.005. Epub 2021 Mar 8. PMID 33705748

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EVO100 | Placebo
Started | 426 | 434
Completed | 335 | 335
Not Completed | 91 | 99
Not completed — Adverse Event | 3 | 3
Not completed — Protocol Violation | 9 | 12
Not completed — Physician Decision | 3 | 6
Not completed — Pregnancy | 7 | 7
Not completed — Withdrawal by Subject | 16 | 22
Not completed — Lost to Follow-up | 37 | 34
Not completed — Other reason not specified | 16 | 15

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- EVO100: A pH-buffering, acidity-maintaining gel (pH 3.5), containing three active compounds: lactic acid, citric acid, potassium bitartrate. 5 g intravaginally applied at least one hour prior to vaginal intercourse.
  EVO100l: 5 g dose applied up to 1 hour prior to coitus
- Total: Total of all reporting groups
Arm/Group | EVO100 | Placebo | Total
Number analyzed (Participants) | 426 | 434 | 860
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 426 | 434 | 860
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.82 (7.112) | 27.53 (6.722) | 27.68 (6.916)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 426 | 434 | 860
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 135 | 148 | 283
  Not Hispanic or Latino | 291 | 286 | 577
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 185 | 173 | 358
  White | 228 | 239 | 467
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 426 | 434 | 860

OUTCOME MEASURES:

1. Primary Outcome: Urogenital CT Infection
Description: Proportion of subjects who experience urogenital CT infection during the study intervention period (incident infection of CT).
Time Frame: 16 weeks
Population: mITT Population - All CT Analysis Eligible Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 289 | 290
Participants | 14 | 28
Statistical Analysis 1: Comparison: EVO100 vs Placebo; Test type: Superiority; p = 0.0256, Chi-squared; Risk Difference (RD) = -4.81, 95% CI 2-sided [-9.02 to -0.61]

2. Secondary Outcome: Urogenital GC Infection
Description: Proportion of subjects who experience urogenital GC infection during the study intervention period (incident infection of GC).
Time Frame: 16 weeks
Population: mITT Population - All GC Analysis Eligible Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 280 | 277
Participants | 2 | 9
Statistical Analysis 1: Comparison: EVO100 vs Placebo; Test type: Superiority; p = 0.0316, Chi-squared; Risk Difference (RD) = -2.53, 95% CI 2-sided [-4.84 to -0.23]

3. Other Pre Specified Outcome: Compliance With EVO100 and Sensitivity Analyses (Part I)
Description: Summary of Coital Events during treatment
Time Frame: 16 weeks
Population: mITT population
Measure: Mean (Standard Deviation); unit: Coital Events
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 364 | 383
Coital Events | 15.7 (14.38) | 16.3 (15.79)

4. Other Pre Specified Outcome: Subject Satisfaction With Product
Description: The proportion of subjects who experienced at least one CT infection during the study Intervention Period was summarized by treatment group using the mITT population and subject adherence rates.
Time Frame: 16 weeks
Population: Subject Satisfaction by Visit (mITT population)
Measure: Count of Participants; unit: Participants
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 273 | 267
Participants
  Very satisfied | 113 | 119
  Satisfied | 128 | 121
  Somewhat Satisfied | 26 | 24
  Somewhat dissatisfied | 5 | 3
  Dissatisfied | 1 | 0

5. Other Pre Specified Outcome: Sexual Satisfaction
Description: The proportion of subjects who experienced at least one GC infection during the study Intervention Period was summarized by treatment group using the mITT population and subject adherence rates.
Time Frame: 16 weeks
Population: Subjects sexual satisfaction by Visit - mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 273 | 267
Participants
  My sex life is a lot better than before | 65 | 53
  My sex life is a little better than before | 75 | 73
  My sex life is no different than before | 124 | 137
  My sex life is a little worse than before | 8 | 4
  My sex life is a lot worse than before | 1 | 0

6. Other Pre Specified Outcome: Compliance With EVO100 and Sensitivity Analyses
Description: as for outcome 4
Time Frame: 16 weeks
Population: mITT Population - All CT Analysis Eligible Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 287 | 290
Participants
  # of subjects w/ CT infection & 0% adherence | 6 | 6
  of subjects w/ CT infection & >0% <20% adherence | 10 | 7
  of subjects w/ CT infection & >=20% adherence | 17 | 13
  of subjects w/ CT infection & >=40% adherence | 19 | 24
  of subjects w/ CT infection & >=60% adhere | 41 | 32
  of subjects w/ CT infection & >=80% adhere | 108 | 125
  of subjects w/ CT infection & =100% adhere | 86 | 83
Statistical Analysis 1: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with =0% adherence; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >0% adherence; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >=20% adherence; Test type: Superiority; p = .6278, Fisher Exact
Statistical Analysis 4: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >=40% adherence; Test type: Superiority; p = .6404, Fisher Exact
Statistical Analysis 5: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >=60% adherence; Test type: Superiority; p = .5008, Fisher Exact
Statistical Analysis 6: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >=80% adherence; Test type: Superiority; p = .1818, Chi-squared
Statistical Analysis 7: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with =100% adherence; Test type: Superiority; p = 0.0012, Chi-squared

7. Other Pre Specified Outcome: Compliance With EVO100 and Sensitivity Analyses
Description: as for outcome 5
Time Frame: 16 weeks
Population: mITT Population - All GC Analysis Eligible Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 279 | 277
Participants
  # of subjects with GC infection & 0% adherence | 5 | 6
  # of subjects w/ GC infection & >0% <20% adherence | 9 | 7
  # of subjects with GC infection & >=20% adherence | 15 | 12
  # of subjects with GC infection & >=40% adherence | 17 | 23
  # of subjects with GC infection & >=60% adh | 40 | 36
  # of subjects with GC infection & >=80% adherence | 106 | 123
  # of subjects with GC infection & =100% adherence | 87 | 70
Statistical Analysis 1: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with =0% adherence; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >0% adherence; Test type: Superiority; p = 0.4375, Fisher Exact
Statistical Analysis 3: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >=20% adherence; Test type: Superiority; p = 0.4444, Fisher Exact
Statistical Analysis 4: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >=60% adherence; Test type: Superiority; p = 0.1836, Fisher Exact
Statistical Analysis 5: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with >=80% adherence; Test type: Superiority; p = 0.5006, Fisher Exact
Statistical Analysis 6: Comparison: EVO100 vs Placebo; A comparison of infection rates between the treatment arms amongst subjects with =100% adherence; Test type: Superiority; p = 1.000, Fisher Exact

8. Other Pre Specified Outcome: Compliance With EVO100 and Sensitivity Analyses (Part II)
Description: Summary of number of applicators used via eDiary
Time Frame: 16 weeks
Population: mITT population
Measure: Mean (Standard Deviation); unit: Number of Applicators
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 360 | 377
Number of Applicators | 13.0 (12.95) | 13.5 (15.18)

9. Other Pre Specified Outcome: Compliance With EVO100 and Sensitivity Analyses (Part III)
Description: Study product adherence
Time Frame: 16 weeks
Population: mITT population
Measure: Mean (Standard Deviation); unit: % of sex acts where study product used
Arm/Group | EVO100 | Placebo
Number analyzed (Participants) | 360 | 377
% of sex acts where study product used | 78.9 (27.14) | 78.3 (27.78)

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: For the 860 subjects randomized into the study, 764 had documented use of study product and were a part of the safety population/analyzed for safety purposes. Amongst these 764 subjects, no deaths were reported during the course of the study.
Arm/Group | EVO100 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/376 | 0/388
Serious Adverse Events (participants affected / at risk) | 2/376 | 3/388
Other Adverse Events (participants affected / at risk) | 62/376 | 46/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVO100 (N=376) | Placebo (N=388)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVO100 (N=376) | Placebo (N=388)
Bacterial Vaginosis (Infections and infestations) | 11 (11) | 18 (18)
Urinary tract infections (Infections and infestations) | 12 (12) | 10 (10)
Vulvovaginal Candidiasis (Infections and infestations) | 19 (19) | 8 (8)
Vaginal Discharge (Reproductive system and breast disorders) | 12 (12) | 10 (10)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 8 (8) | 0 (0)

LIMITATIONS AND CAVEATS:
For the Adverse Event Section: There were no All-Cause Mortalities to Report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT03107377/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03107377/SAP_001.pdf